CLINICAL TRIAL: NCT05918952
Title: RADx-UP CDCC Rapid Research Pilot Program: "Culturally-relevant Community Connections (C3) to Increase COVID-19 Testing in the Black/African American Community".
Brief Title: RADx-UP CDCC Rapid Research Pilot Program "Culturally-relevant Community Connections (C3) to Increase COVID-19 Testing
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00112394; R0606A (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2023-06-21; First posted 2023-06-26 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Covid-19 antibody test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Culturally-relevant Community Connections (C3): 1-health COVID-19 test and Video
  Interventions: Diagnostic Test: Covid-19 Antibody Test; Other: Short Clip videos

INTERVENTIONS:
Diagnostic Test: Covid-19 Antibody Test — The investigators propose to use the iHealth® Rapid COVID-19 Antigen Rapid Test. Per the EUA guidance, study participants will complete one test at a study location and receive one test to take home with instructions to complete it within 48 hours.
  Each testing site will have a private designated space for customers to self-collect and test themselves privately. The edutainment video will serve as a resource for information on accurate test performance. Test one will be done in a private setting and results entered into REDcap and will also be written on a testing card with contact information for the purpose of follow-up. For test number two the customer will self-collect within 48 hours (per the FDA EUA for this particular test) and results will be entered into RedCap.
Other: Short Clip videos — Designed to discuss the testing process, the importance of getting tested and accessing care, and how COVID-19 has disproportionately affected the Black/African-American community.

SUMMARY:
The purpose of this study is to identify barriers and facilitators to COVID testing among members of the Black/African American community. The expected outcome of this project is to increase COVID testing among Black/African American community. The secondary aim is to examine the use of culturally relevant edutainment video messaging combined with trusted opinion leaders in the community as a strategy to increase COVID testing.

DETAILED DESCRIPTION:
The pandemics of COVID-19 and racial discrimination in America have joined forces to illuminate inequalities in healthcare delivery and health outcomes of Black Americans. These pandemics have increased attention to the medical distrust, racism, discrimination, implicit bias, and unequal treatment that has occurred in this country for centuries.

Trusted venues such as barber shops and beauty salons are gatekeepers and facilitators of trusted information in the Black community. The investigators are addressing Health disparities through Engagement, Equity, Advocacy, and Trust (HEEAT) Research Lab partners with barbers and stylists for health promotion in communities of color. The investigators co-founded North Carolina Barbers and Stylists for Health Equity (NCBSHE), a network of barber shops and beauty salons serving primarily Black clientele throughout NC. NCBSHE is led by barbers and stylists, with academic partners serving the organization in non-leadership roles.

Due to barriers including access to care, discrimination, and medical distrust, engaging the Black community in health research and improvement activities requires a community-based approach. The investigators' novel approach integrates evidence-based strategies that will address these barriers to engagement. The success of this project in increasing the uptake of COVID-19 testing in the Black community will serve as a model for other health-related activities beyond COVID.

Research Approach

The investigators' current and prior work addressing HIV prevention among Black women successfully trained stylists in the community to bring awareness and knowledge of pre-exposure prophylaxis (PrEP). The first three months of this COVID-19 project will focus on training stylists and barbers as Opinion Leaders (OLs), development of edutainment videos, and training of research staff. An NP will provide telehealth support to customers who test positive, and the Community Coordinator will facilitate the OL workshop. The workshop will include updates on COVID-19 in the designated testing areas, CDC guidelines for COVID-19, clinical presentation, prevention strategies, testing, and telehealth policies and procedures, and roles and responsibilities of an OL. An OL serves as a community liaison between the researcher and the community. They do not serve as interventionists but are informed of research practices and current studies taking place in their community.

Investigators will partner with an established communication strategist team we have previously worked with to co-develop culturally and socially relevant short clip edutainment videos.

OLs training as an evidence-based model to promote health. Without ready and convenient access to credible, peer-reviewed information, people in search of information about health and well-being appear to turn to trusted local information sources such as personal connections and trusted healthcare professionals. Kim and colleagues note the importance of social networks and local information sources among underserved communities. Training of beauty industry professionals as OLs has been promising. There is evidence that customer confidence is increased when stylists undertake workshops in preparation for sharing information.

Edutainment videos are an evidence-based intervention strategy for health promotion and prevention among communities of color. Grounded in transportation theory, edutainment videos are designed to entertain and improve literacy while communicating prosocial norms and behaviors. These short clip videos will be accessible by scanning a QR code in the barber shop or beauty salon. A trained beauty professional will offer each client the opportunity to view the video. A $5 off coupon for hair services with the designated salon/shop will be offered if the client watches the video. At the end of the video, the client will be asked if they would like to be tested that day. If they respond no, the client will be asked a set of questions that explain the reason (e.g., I was tested in the past 2 weeks, I prefer to get tested at my doctor's office, I don't think I have COVID, I don't trust the COVID test). If the customer says yes, the client will be asked a set of questions about the reason for the decision (facilitators) (e.g., I feel comfortable testing in this space, the video encouraged me to be tested today, I have been wanting to get tested, but did not have easy access to testing).

A nurse-led model of care: the role of the advanced practice nurse and telehealth. NPs are positioned to advance health equity and support efforts to improve testing in the community. In prior work by the team and others, the nursing workforce is increasingly being recognized as being uniquely positioned to drive healthcare innovation to advance health equity. A recent National Academies of Sciences, Engineering, and Medicine (NASEM) report outlined a comprehensive vision for nurse-led innovation as a driving force in overhauling conventional models of health service delivery. Specifically, the NASEM report endorses the scale-up of nurse-led interdisciplinary care delivered directly in community settings. The NP will be a liaison for OLs and salons/shops and will contact customers who test positive for COVID to educate them of next steps. Since COVID, telehealth has been used to improve access to care and address barriers such as transportation, childcare limitations, and needing time off for appointments. Telehealth addresses traditional barriers to and disparities in access to care while also improving efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black/African American
* 18 Years and older
* visit the beauty salon or barber shop to enroll in the study

Exclusion Criteria:

* under the age of 18
* non Black/African American identifying

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black/African American adults
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schenita Randolph, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Hair Designs By Tasha, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two beauty salons and three barbershops agreed to partner to implement this project. Recruitment of customers in these shops took place through word of mouth, an IRB-approved recruitment flyer, and through the co-developed edutainment videos.
Groups:
- Culturally-relevant Community Connections (C3): 1-health COVID-19 test and Video
  Covid-19 Antibody Test: The investigators propose to use the iHealth® Rapid COVID-19 Antigen Rapid Test. Per the EUA guidance, study participants will complete one test at a study location and receive one test to take home with instructions to complete it within 48 hours.
  Each testing site will have a private designated space for customers to self-collect and test themselves privately. The edutainment video will serve as a resource for information on accurate test performance. Test one will be done in a private setting and results entered into REDcap and will also be written on a testing card with contact information for the purpose of follow-up. For test number two the customer will self-collect within 48 hours (per the FDA EUA for this particular test) and results will be entered into RedCap.
  Short Clip videos: Designed to discuss the testing process, the importance of getting tested and accessing care, and how COVID-19 has disproportionately affected the Black/African-American community.
Period: Overall Study
Arm/Group | Culturally-relevant Community Connections (C3)
Started | 327
Completed | 327
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Culturally-relevant Community Connections (C3)
Number analyzed (Participants) | 327
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.26 (13.32)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 186
  Sex/Gender: Male | 128
  Sex/Gender: Other | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 310
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 315
  White | 0
  More than one race | 12
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completed COVID-19 Tests
Time Frame: 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally-relevant Community Connections (C3)
Number analyzed (Participants) | 327
Participants | 73
Statistical Analysis 1: Comparison: Culturally-relevant Community Connections (C3); Test type: Superiority; p = .05, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.21 to 3.98]

2. Primary Outcome: COVID-19 Testing Decision-Making Scale (CTDMS) General Sentiment (GS) Subscale
Description: The CTDMS is an 8-item measure with 2 subscales: General Sentiment (4 items) and Practical Support (4 items). The GS subscale score is calculated as a mean with a range of 1 to 5. Higher scores indicate stronger agreement with positive general attitudes and experiences toward COVID-19.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Culturally-relevant Community Connections (C3)
Number analyzed (Participants) | 327
score on a scale | 2.41 (0.93)
Statistical Analysis 1: Comparison: Culturally-relevant Community Connections (C3); Hypothesis: Higher General Sentiment (GS) scores will be associated with greater likelihood of COVID-19 testing uptake; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.35 to 2.41]

3. Secondary Outcome: Video Feedback Scale (VFS)
Description: The VFS contains 9 items, each with a response scale of 1 to 5. The VFS total score is calculated as a mean with a range of 1 to 5. Higher scores indicate greater perceived impact, cultural resonance, and acceptability of the intervention videos for health behavior change.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally-relevant Community Connections (C3)
Number analyzed (Participants) | 327
units on a scale | 4.27 (0.64)
Statistical Analysis 1: Comparison: Culturally-relevant Community Connections (C3); Hypothesis: Higher VFS scores will be associated with increased likelihood of test uptake; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.54, 95% CI 2-sided [2.01 to 6.20]
Statistical Analysis 2: Comparison: Culturally-relevant Community Connections (C3); Hypothesis: Higher VFS scores will be associated with increased likelihood of completion of a follow-up test; Test type: Other; p = 0.029, Regression, Logistic — Low sample size and power. Model considered unstable and potentially overfit. Results not reliable; Odds Ratio (OR) = 11.01, 95% CI 2-sided [1.27 to 95.17]

4. Primary Outcome: COVID-19 Testing Decision-Making Scale (CTDMS) Practical Support (PS) Subscale
Description: The CTDMS is an 8-item measure with 2 subscales: General Sentiment (4 items) and Practical Support (4 items). The PS subscale score is calculated as a mean with a range of 1 to 5. Higher scores reflect greater perceived practical support for testing (e.g., importance, accessibility).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Culturally-relevant Community Connections (C3)
Number analyzed (Participants) | 327
score on a scale | 3.68 (0.80)
Statistical Analysis 1: Comparison: Culturally-relevant Community Connections (C3); Hypothesis: Higher Practical Support (PS) scores will be associated with greater likelihood of COVID-19 testing uptake; Test type: Other; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.19 to 2.40]

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Groups:
- Testing Group: 1-health COVID-19 test and Video
  Covid-19 Antibody Test: The investigators propose to use the iHealth® Rapid COVID-19 Antigen Rapid Test. Per the EUA guidance, study participants will complete one test at a study location and receive one test to take home with instructions to complete it within 48 hours.
  Each testing site will have a private designated space for customers to self-collect and test themselves privately. The edutainment video will serve as a resource for information on accurate test performance. Test one will be done in a private setting and results entered into REDcap and will also be written on a testing card with contact information for the purpose of follow-up. For test number two the customer will self-collect within 48 hours (per the FDA EUA for this particular test) and results will be entered into RedCap.
  Short Clip videos: Designed to discuss the testing process, the importance of getting tested and accessing care, and how COVID-19 has disproportionately affected the Black/African-American community.
Arm/Group | Testing Group
All-Cause Mortality (participants affected / at risk) | 0/327
Serious Adverse Events (participants affected / at risk) | 0/327
Other Adverse Events (participants affected / at risk) | 0/327

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT05918952/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT05918952/ICF_000.pdf